CLINICAL TRIAL: NCT03318757
Title: Does Bupivacaine Liposomal Injectable Suspension Decrease Post-operative Pain and Narcotic Use After Elective Orthognathic Surgery?
Brief Title: Bupivacaine Liposomal Injectable Suspension, Pain and Narcotic Use After Elective Orthognathic Surgery
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The research could not be conducted as it was denied by the IRB.
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-36862
Record Dates: First submitted 2017-10-15; First posted 2017-10-24 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Orthognathic Surgery
Keywords: bupivacaine liposomal injectable; post operative pain; post operative narcotic use; bupivacaine hydrochloride
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1- Bupivacaine extended release liposome injection (Experimental): Bupivacaine extended release liposome injection (Exparel TM) is a novel formulation of bupivacaine designed to achieve long-acting postoperative analgesia.
  Interventions: Drug: Bupivacaine Extended Release Liposome Injection
- Group 2- Bupivacaine HCl (Active Comparator): Bupivacaine HCl (Marcaine) is a local anesthetic that reduces the flow of sodium in and out of nerves which decreases the initiation and transfer of nerve signals in the area in which the drug is applied.
  Interventions: Drug: Bupivacaine HCl

INTERVENTIONS:
Drug: Bupivacaine Extended Release Liposome Injection — Bupivacaine Extended Release Liposome Injection (Exparel TM) 133 mg diluted in 10ml of normal saline (13.3 mg/ml) will be injected with a 25 gauge needle directly into the gingiva surrounding the surgical site at the conclusion of surgery.
  Other Names: Exparel TM
  Arms: Group 1- Bupivacaine extended release liposome injection
Drug: Bupivacaine HCl — 10ml of Bupivacaine HCl 0.5% will be injected with a 25 gauge needle directly into the gingiva surrounding the surgical site at the conclusion of surgery.
  Other Names: Marcaine
  Arms: Group 2- Bupivacaine HCl

SUMMARY:
This research is being done to determine quantitative and qualitative differences in patients' post-operative pain levels following elective orthognathic surgery after the local administration of a liposomal bupivacaine injection.

A primary objective is to determine whether using a liposomal bupivacaine injection placed locally at the conclusion of elective orthognathic surgery will decrease pain levels (as determined by VAS scores). A secondary objective is to examine whether using a long acting liposomal bupivacaine injection locally at the conclusion of elective orthognathic surgery leads to decreased use of narcotics post-operatively.

DETAILED DESCRIPTION:
Participants in Group 1 (study group) will receive ExparelTM (133 mg/10 ml - 4 ml into the maxilla, and 6 ml into the mandible). This will be injected into the soft tissue and gingiva surrounding the surgical site at the time of wound closure. Participants in Group 2 (standard of care) will receive bupivacaine 0.5% (4 ml into the maxilla, and 6 ml into the mandible) injected into the soft tissue and gingiva surrounding the surgical site at the time of wound closure.

Post-operatively, all participants will be cared for utilizing the current standard post-operative pain management protocol for all patients undergoing elective orthognathic surgery at Boston Medical Center. This consists of acetaminophen 325 mg given every 4 hours as a scheduled medication; patients also receive an additional 325 mg of acetaminophen for a reported pain level of 1-3, 5 mg of oxycodone for a reported pain level of 4-6, and 10 mg of oxycodone for a reported pain level of 7-10. All participants will be provided the same methods of postoperative pain control following their elective orthognathic surgery.

ELIGIBILITY:
Inclusion Criteria:

* males and females 18-40 years of age undergoing elective double jaw orthognathic surgery

Exclusion Criteria:

* pregnancy
* known hypersensitivity to any local anesthetic

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in Post operative pain | 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 72, and 96 hours after surgery
  After surgery, participants will document in a pain journal what their pain level is based on a smiley face visual analog scale (VAS) from 0-10, where 0='no pain' and 10='worst possible, unbearable, excruciating pain'. They will rate their pain using the VAS 14 times - every 4 hours the first 48 hours and then at 72 and 96 hours post surgery. Higher scores are associated with more severe pain. The participant will return the pain journal at their post operative assessment visit.

SECONDARY OUTCOMES:
Post operative narcotic use | daily up to the 2 week post surgical visit
  The time and dosage of narcotics used in the postoperative period will be documented in the participants' medical record records while hospitalized and documented in the participants' pain journal once discharged. The data from the medical records and pain journal will be used to assess total narcotic pain use.

CONTACTS AND LOCATIONS:
Overall Officials: Pushkar Mehra, BDS DMD, Principal Investigator — BU Henry M. Goldman School of Dental Medicine
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No